CLINICAL TRIAL: NCT01396772
Title: A Community-based Healthy Lifestyle Patient-centred Education Program for Middle & Older Adults With Prediabetes, Which Strengthens the Delivery of Health Services and Assists Individuals at High-risk for Diabetes in London, Ontario.
Brief Title: PREPARE: "Prediabetes Research and Education Promoting Activity & Responsible Eating"
Acronym: PREPARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brescia University College (Other)
Responsible Party: Isabelle Giroux, Ph.D., R.D., B.Ed., P.H.Ec., Associate Professor, Brescia University College, affiliated with The University of Western Ontario
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRT-2010-012
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Prediabetes
Keywords: prediabetes; diabetes prevention; adults; lifestyle intervention; Social Cognitive Theory; dietary intake; physical activity
MeSH Terms: conditions — Prediabetic State; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PREPARE education program (Experimental): This is a 6-month program that consists of monthly nutrition and physical activity education sessions (2 hours per session) and includes interactive hands-on activities to help you gain knowledge and skills to make positive lifestyle choices. It is a pilot study to test the effectiveness of this type of health-care program in individuals with prediabetes.
  Interventions: Behavioral: PREPARE education program
- Control arm (Other): Individuals self-selecting the control arm receive the current standard of care for prediabetes, which is a one-time 2-hour group education session. In addition, the individuals are asked to provide some information at baseline and 6 months and 1 year later. The information collected will include a record of dietary and physical activity habits and whether or not they have developed Type 2 diabetes.
  Interventions: Other: standard of care presentation

INTERVENTIONS:
Behavioral: PREPARE education program — PREPARE stands for "Prediabetes Research and Education Promoting Activity and Responsible Eating" and is a 6-month community-based prediabetes lifestyle and behaviour change intervention program. It includes a series of six interactive education sessions of two hours each on healthy eating and physical activity.
  Other Names: Prediabetes Research and Education Program
  Arms: PREPARE education program
Other: standard of care presentation — A one-time 2-hour group prediabetes education session, offered as the standard for individuals referred for prediabetes in London, Ontario (Canada)
  Other Names: Standard
  Arms: Control arm

SUMMARY:
The purpose of this study is to determine if a 6-month community-based prediabetes lifestyle and behaviour change intervention (called, PREPARE) for middle and older adults with prediabetes will result in positive lifestyle behaviour change.

DETAILED DESCRIPTION:
This community-based, healthy lifestyle project targets middle (30-59) and older (60+) adults with prediabetes - a population known to be at high risk for Type 2 diabetes development.

This project aims to create, deliver and evaluate a six month interdisciplinary education and lifestyle improvement intervention that emphasizes goal-setting and self-management approaches to inform, engage, monitor and support adults with prediabetes in making positive lifestyle changes within the London (Ontario, Canada) community.

Participants are encouraged to reflect on their current lifestyle, resources and barriers, increase skills, motivation, and awareness of community resources, and make positive lifestyle changes. Based on a solid partnership between both community - health service providers and Brescia University College, the Prediabetes Initiative aims at empowering individuals with prediabetes through self-management approaches to reduce behaviours known to contribute to Type 2 diabetes development.

ELIGIBILITY:
Inclusion Criteria:

* Adults; 30 years of age or older, residing in the London (Ontario, Canada) or surrounding area (including Middlesex), who currently have prediabetes diagnosed by their health care provider (e.g. family physician) and who have been referred to the Diabetes Education Centre of St. Joseph's Health Care London by a physician.
* Eligible participants must not be currently participating in another lifestyle or behaviour change education or research program; must be able to perform low impact physical activity; must be able to eat a balanced diet; must not be lactating or pregnant; and must be able to understand English enough to participate in the educational discussions and activities and to fill in required questionnaires.
* Eligible participants must not be diagnosed with Type 1 or Type 2 diabetes, or any condition (e.g. cancer, etc) or behavioural or psychiatric issues (such as a diagnosis of major depression, eating disorder, schizophrenia or other mental illness) as this will prevent full engagement in the program.

Exclusion Criteria:

* Non-adults; adults of less than 30 years of age; adults residing outside the London (Ontario, Canada) and surrounding area; adults who do not currently have a diagnosis of prediabetes and have not been referred to the Diabetes Education Centre of St. Joseph's Health Care London by a physician
* Individuals currently participating in another lifestyle or behaviour change education or research program.
* Not being able to perform low impact physical activity, such as being chair-bound or having low mobility;
* Being unable to chew and digest food normally and to eat a balanced diet (e.g. being on a specialized diet such as a low-fiber diet or enteral nutrition support due to a pre-existing condition, such as Crohn's disease, celiac disease or other digestive disease);
* Currently lactating or being pregnant;
* Being unable to understand, read and write the English language; or
* Having a diagnosis of Type 1 or Type 2 diabetes, or any condition (e.g. cancer, etc) or behavioural or psychiatric issues (such as a diagnosis of major depression, anorexia nervosa, bulimia nervosa, eating disorder not otherwise specified [EDNOS], schizophrenia or other mental illness) that would prevent full engagement in the program.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Average number of vegetable and fruit servings consumed per day | Baseline, 6 months and 12 months after the baseline assessment
  Data collected using a standard 3-Day Food Intake Record and Medication Log form at the three time points.

SECONDARY OUTCOMES:
average number of physical activity minutes per day | Baseline, 6 months and 12 months after the baseline assessment
  Data collected using a 7-Day Physical Activity and Step Log standard form.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle T. Giroux, PhD, Principal Investigator — Brescia University College
Locations (1):
- Brescia University College, London, Ontario, Canada

REFERENCES:
- See also: Prediabetes Initiative and Partnership — http://www.brescia.uwo.ca/prediabetes_initiative/